CLINICAL TRIAL: NCT04475926
Title: Journey: A Global, Multicenter, Longitudinal Study of the Natural History of Subjects With Limb Girdle Muscular Dystrophy (LGMD) Type 2E (LGMD2E/R4), Type 2D (LGMD2D/R3), Type 2C (LGMD2C/R5), and Type 2A (LGMD2A/R1)
Brief Title: A Study of the Natural History of Participants With LGMD2E/R4, LGMD2D/R3, LGMD2C/R5, and LGMD2A/R1 ≥ 4 Years of Age, Who Are Managed in Routine Clinical Practice
Status: Active, not recruiting | Type: Observational
Sponsor: Sarepta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SRP-LGMD-501-NHS
Record Dates: First submitted 2020-07-14; First posted 2020-07-17 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Limb-girdle Muscular Dystrophy
Keywords: North Star Assessment for Dysferlinopathy (NSAD); Performance of Upper Limb (PUL); Pulmonary function tests (PFTs); Ambulatory; Non-Ambulatory; Limb-girdle; LGMD; sarcoglycanopathy; β -sarcoglycan; Muscular Dystrophy; α -sarcoglycan; γ -sarcoglycan; LGMD-2D/R3; LGMD-2E/R4; LGMD-2C/R5; LGMD2A/R1; Clinical Outcomes Assessment
MeSH Terms: conditions — Muscular Dystrophies, Limb-Girdle; Sarcoglycanopathies; Muscular Dystrophies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (4):
- LGMD2E/R4 Cohort: Participants with LGMD2E/R4 will be enrolled in this cohort. Enrollment will be capped according to age as follows: 4 to 7 years age range, 8 to 16 years age range, and ≥17 years age range through the course of the study.
- LGMD2D/R3 Cohort: Participants with LGMD2D/R3 will be enrolled in this cohort. Enrollment will be capped according to age as follows: 4 to 7 years age range, 8 to 16 years age range, and ≥17 years age range through the course of the study.
- LGMD2C/R5 Cohort: Participants with LGMD2C/R5 will be enrolled in this cohort. Enrollment will be capped according to age as follows: 4 to 7 years age range, 8 to 16 years age range, and ≥17 years age range through the course of the study.
- LGMD2A/R1 Cohort: Participants with LGMD2A/R1 will be enrolled in this cohort. Enrollment will be capped according to age as follows: 4 to 7 years age range, 8 to 16 years age range, and ≥17 years age range through the course of the study.

SUMMARY:
This study will follow participants who are screened and confirmed with a genetic diagnosis of Limb-girdle muscular dystrophy type 2E (LGMD2E/R4), Limb-girdle muscular dystrophy type 2D (LGMD2D/R3), Limb-girdle muscular dystrophy type 2C (LGMD2C/R5), or Limb-girdle muscular dystrophy type 2A (LGMD2A/R1).

These enrolled participants will be followed to evaluate mobility and pulmonary function for up to 5 years after enrollment for participants with LGMD2C/R5, LGMD2D/R3, and LGMD2E/R4 with a North Star Assessment for Dysferlinopathy (NSAD) ≥ 25 at Baseline, up to 3 years for participants with LGMD2C/R5, LGMD2D/R3, and LGMD2E/R4 with a NSAD < 25 at Baseline, and up to 3 years for participants with LGMD2A/R1. Additional participant data will be collected from the time the individual began experiencing LGMD symptoms to the present.

DETAILED DESCRIPTION:
LGMD Type 2A, 2C, and 2D cohorts are now closed. Enrollment in the LGMD Type 2E cohort is closed and participants will be followed for up to five years.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participant ≥ 4 years of age who demonstrate symptoms of LGMD2E/R4, LGMD2D/R3, LGMD2C/R5, or LGMD2A/R1 in the opinion of the investigator (eg, muscle weakness, loss of function, delayed milestones).
* Confirmed clinical and genetic diagnosis of LGMD2E/R4, LGMD2D/R3, LGMD2C/R5, or LGMD2A/R1.

Exclusion Criteria:

* Demonstrates cognitive delay or impairment that could confound motor development, in the opinion of the Investigator.
* Has a medical condition, in the opinion of the Investigator, that might compromise participants ability to comply with study requirements.
* Is participating in other interventional study(ies) at the time of enrollment in this study.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population for this study is ambulatory or non-ambulatory participants ≥ 4 years of age with confirmed genetic diagnosis of LGMD2E/R4, LGMD2D/R3, LGMD2C/R5, or LGMD2A/R1.
Sampling Method: Non-Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2030-09-05 (Estimated); Study Completion 2030-09-05 (Estimated)

PRIMARY OUTCOMES:
NSAD Total Score | Baseline up to Month 60
Time to Rise from the Floor | Baseline up to Month 60
Time of 10-Meter Walk/Run [10MWR] | Baseline up to Month 60
Time to Ascend 4 Steps | Baseline up to Month 60
Ankle Range of Motion (ROM) | Baseline up to Month 60
Dimension of the Performance of the Upper Limb (PUL) | Baseline up to Month 60
Timed Up and Go (TUG) | Baseline up to Month 60
Time of 100-Meter Walk/Run (100MWR) | Baseline up to Month 60
Pulmonary Function Test: Forced Vital Capacity (FVC) | Baseline up to Month 60

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sarepta Therapeutics, Inc.
Locations (26):
- United States (11):
  - Barrow Neurological Institute, Phoenix, Arizona
  - Arkansas Children's, Little Rock, Arkansas
  - University of California San Diego, La Jolla, California
  - University of California, Davis Health Dept of PM&R, Sacramento, California
  - Anne & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Utah Hospital, Salt Lake City, Utah
  - Children's Hospital of the King's Daughters, Norfolk, Virginia
- Belgium (3):
  - University Hospital Gent, Ghent, Oost-Vlaanderen
  - UZ Leuven, Leuven, Vlaams Brabant
  - Hôpital Universitaire des Enfants Reine Fabiola, Brussels
- Hospital de Clinicas de Porto Alegre (HCPA) - PPDS, Porto Alegre, Rio Grande do Sul, Brazil
- Children's Hospital - London Health Science Centre, London, Ontario, Canada
- Germany (2):
  - Zentrum für Kinderheilkunde und Jugendmedizin Uniklinikum Giessen Marburg (UKGM), Standort Giessen, Giessen, Hesse
  - Universitätsklinikum Essen, Essen, North Rhine-Westphalia
- Italy (3):
  - Istituto Giannina Gaslini, Genoa, Liguria
  - Azienda Ospedale Università Padova, Padua, Veneto
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
- Hospital Sant Joan de Déu Universidad de Barcelona, Barcelona, Spain
- Karolinska Universitetssjukhuset Solna, Stockholm, Stockholm County, Sweden
- Lokman Hekim Etlik Hastanesi, Ankara, Turkey (Türkiye)
- United Kingdom (2):
  - UCL Institute of Child Health & Great Ormond Street Hospital for Children, London
  - Institute of Genetic Medicine, International Centre for Life, Newcastle upon Tyne